CLINICAL TRIAL: NCT04061655
Title: Effect of Intravenous Iron Supplementation in Reducing Allogenic Blood Transfusion and Improving Outcomes in Patients Undergoing CABG. A Prospective Randomized Trial
Brief Title: Effect of Intravenous Iron Supplementation in Reducing Allogenic Blood Transfusion
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Hoda Shokri, Associate professor of Anesthesia, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: FMASU R 03/ 2019
Record Dates: First submitted 2019-08-17; First posted 2019-08-20 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Complications
Keywords: CABG; iron therapy; blood transfusion
MeSH Terms: interventions — iron isomaltoside 1000

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- iron therapy group (Active Comparator): Apatients (n= 40) received single dose intravenous infusions of iron isomaltoside 1000 mg over 15 min with a maximum single dose of 20 mg/kg.
  Interventions: Drug: Iron Isomaltoside 1000
- placebo (Placebo Comparator): Patients in the placebo group (n=40)received as a single-dose of saline (Natriumklorid 9 mg/ml; Fresenius Kabi, Copenhagen, Denmark) 100 ml infused over 15 min.
  Interventions: Other: placebo

INTERVENTIONS:
Drug: Iron Isomaltoside 1000 — Apatients (n= 40) received single dose intravenous infusions of iron isomaltoside 1000 mg over 15 min with a maximum single dose of 20 mg/kg.
  Other Names: iron therapy
  Arms: iron therapy group
Other: placebo — Patients in the placebo group (n=40)received as a single-dose of saline (Natriumklorid 9 mg/ml; Fresenius Kabi, Copenhagen, Denmark) 100 ml infused over 15 min.
  Arms: placebo

SUMMARY:
A total of 80 patients will be randomly allocated into 2 groups, group A and placebo group using concealed envelope method.Group A patients (n= 40)will receive single dose intravenous infusions of iron isomaltoside 1000 mg over 15 min with a maximum single dose of 20 mg/kg. Patients in the placebo group (n=40) will receive as a single-dose of saline (Natriumklorid 9 mg/ml; Fresenius Kabi, Copenhagen, Denmark) 100 ml infused over 15 min.

DETAILED DESCRIPTION:
A total of 80 patients will randomly allocated into 2 groups, group A and placebo group using concealed envelope method.Group A patients (n= 40) will receive single dose intravenous infusions of iron isomaltoside 1000 mg over 15 min with a maximum single dose of 20 mg/kg. Patients in the placebo group (n=40) will receive as a single-dose of saline (Natriumklorid 9 mg/ml; Fresenius Kabi, Copenhagen, Denmark) 100 ml infused over 15 min.

General anesthesia will the institutional standards and all surgeries will be performed by the same surgical team.Standardized monitoring will be applied.After median sternotomy,CPB will be established with 1500 ml crystalloid priming volume and mild hypothermia (32°C) with a Trillium Affinity oxygenator (Medtronic,Minneapolis, Minnesota, USA) and a Sarns CPB machine (Harrison, Mt. Clemens, Michigan, USA) at a flow rate of 2.6 lmin-1m-2.Myocardial protection will be done using cold blood cardioplegia at 20°C. During CPB, homologous donor packed red blood cells will be transfused if hemoglobin was less than 6.5 gdl-1.During bypass, anticoagulation for extracorporeal circulation was performed using heparin 300 U/kg administered into the right atrium. Acelite activated clotting time (ACT) greater than 400 was considered adequate for commencing CPB; if less, an additional dose of 100Uof heparin will be adminstered.CPB will be conducted using nonocclusive roller pumps, arterial line filtration ,membrane oxygenators, , and blood-enriched cold hyperkalemic arrest. Systemic hypothermia documented by an esophageal temperature of 32°C will be maintained during aortic cross clamping.After completion of CPB and removal of the arterial cannula, heparin will be neutralized with 1 mg of protamine sulfate adminstered for every 100U of heparin over a period of 15 minutes . Eventually, a second dose of protamine 50 mg will be given if ACT remained above baseline. All patients will be transferred to ICU after surgery.

ELIGIBILITY:
Inclusion Criteria:

* patients aged 52-73 years old
* ASA II/III
* elective CABG
* hemoglobin level at baseline for males >13.0 g/dl and for females >12.0 g/dl.

Exclusion Criteria:

* Patients with known hypersensitivity to iron sucrose
* history of hepatitis B or C or human immunodeficiency virus
* folate or vitamin B12deficiency, history of unstable angina,
* active severe infection
* suspicion of iron overload (ferritin > 300 μg/l ), or autologous blood transfusion in the previous month pregnancy and nursing impaired renal function defined by s-creatinine >150 μmol/L patients received any iron preparations in the previous month -

Ages: 52 Years to 73 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2019-09-20 (Actual); Primary Completion 2020-01-06 (Actual); Study Completion 2020-01-10 (Actual)

PRIMARY OUTCOMES:
haemoglobin concentration change | 1 week after discharge from hospital
  the change in the Hb concentration at baseline, intraoperative, at discharge and 1 week after discharge in non-anaemic patients undergoing cardiac surgery.

SECONDARY OUTCOMES:
hospital stay | 7 to 10 days
  duration of hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Ayman Shoeb, professor, Study Director — Ain Shams University
Locations (1):
- Ain Shams university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
study protocol statistical analysis data analysis
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 6 months
Access Criteria: Descriptive statistics will be carried out for numerical parametric data and presented as mean±SD, whereas categorical data will be presented as number and percentage. Variables such as demographic data and comorbidities will be compared using the χ2-test